CLINICAL TRIAL: NCT05619757
Title: Compliance With Medical Treatment for Endometriosis : a Cross-sectional Study
Brief Title: Compliance and Endometriosis
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0547
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pain; Drug treatments; Hormonal treatment; Compliance; Amenorrhea; Recommendations; Menstruation; Quality of life; Efficiency
MeSH Terms: conditions — Endometriosis; Pain; Patient Compliance; Amenorrhea | interventions — Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Compliance with medical treatment for endometriosis — During their scheduled consultation at the Hôpital Femme Mère Enfant (HFME), women who meet the eligibility criteria will be presented with the study and given the written information note. If they agree to participate, the investigator will give them a QR code redirecting them to the online self-questionnaire.
  Patients will be included once they log in and complete the questionnaire.

SUMMARY:
Endometriosis is defined as the presence of hormone-dependent endometrial tissue outside the uterine cavity. It is a chronic, painful and often disabling pathology during the normal activities of daily life. It affects 10% of women of childbearing age. It is therefore a real public health issue.

The latest recommendations from the HAS and the CNGOF now recommend primary medical management of endometriosis in painful women who do not wish to become pregnant. It should be remembered that until very recently, the teams resigned themselves to carrying out surgical interventions in order to support the diagnosis (this is histological and requires a biopsy) and to treat the patient if possible. Sometimes, this treatment was not possible from the outset, as the lesions appeared to be inaccessible, and additional hormonal treatment was therefore required. The current concept is to propose to patients a first hormonal suppressive treatment before a possible surgery. This therapeutic de-escalation should be considered in the light of the physiopathology of endometriosis, which is essentially based on the ovarian cycles, and indirectly on menstruation, which must then be suspended. However, a good number of patients are initially reluctant to undergo any kind of hormonal therapy, either because they have had a bad experience with hormonal contraception (intolerance) or because of a fear related to the possible complications of hormonal therapy with third or fourth generation pills, for example (thromboembolic risk). There is also a health alert at present concerning macro progestins in relation to the risk of meningioma. Acceptance of the principle of instituting amenorrhea in order to relieve patients suffering from endometriosis requires prior information. In investigator's daily practice, they frequently deplore non-compliance, which is detrimental to the proper management of the disease. The effectiveness of hormonal treatment, which will institute a quiescence of hormonal activity, is not immediate. An analgesic and anti-inflammatory treatment is then added. Investigators propose to compare the compliance of three drug strategies: analgesics alone, hormone therapy alone or hormone therapy and analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman with diagnosed painful endometriosis
* Have a prescription for medication (analgesics alone, hormone therapy alone or hormone therapy and analgesics).
* Speak and understand French
* Be a woman over 18 years old until menopause
* Agree to participate in the study

Exclusion Criteria:

- Be a woman who has already had surgery for endometriosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include women with painful endometriosis who have never had endometriosis surgery. In addition, patients must speak and understand French and be over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Compliance measured by the Morisky Medication Adherence Scales (MMAS-8). | 10 minutes
  This self-administered questionnaire validated in French has 8 items each scored 0 or 1. A high score indicates high compliance: high compliance (score = 8), average compliance (score of 6 to < 8) and low compliance (score < 6). Patients with a score greater than or equal to 6 will be considered as compliant. This questionnaire has been validated in French.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie-Obstétrique, Sénologie et Oncologie, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No